CLINICAL TRIAL: NCT05330312
Title: A Randomized, Controlled, Parallel-group Clinical Investigation Evaluating the Impact of Digital Cognitive Behavioural Therapy on Psychological Symptom Burden in Adults Diagnosed With Pulmonary Fibrosis
Brief Title: Controlled Investigation to Evaluate Impact of dCBT on Psychological Symptom Burden in Adult Subjects With PF
Acronym: COMPANION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vicore Pharma AB (Industry)
Collaborators: Curebase Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VP-dCBT-PF-101
Record Dates: First submitted 2022-03-03; First posted 2022-04-15 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Pulmonary Fibrosis; Anxiety
MeSH Terms: conditions — Pulmonary Fibrosis; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The investigation consisted of a Part 1 (pilot phase) with a single arm (4 weeks of dCBT), and a Part 2 (pivotal phase) with a randomised, controlled, parallel-group design to either 9 weeks of dCBT or a control group with no intervention.
Who Masked: Outcomes Assessor
Masking Description: HAM-A raters are blinded (HAM-A = Hamilton Anxiety Rating Scale).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Part 1 - Digital cognitive behavioral therapy (Experimental): 4 weeks digital cognitive behavioral therapy.
  Interventions: Device: Digital cognitive behavioral therapy
- Part 2 - Control group (No Intervention): No intervention
- Part 2 - Digital cognitive behavioral therapy (Experimental): 9 weeks digital cognitive behavioral therapy
  Interventions: Device: Digital cognitive behavioral therapy

INTERVENTIONS:
Device: Digital cognitive behavioral therapy — Therapy for patients with pulmonary fibrosis
  Other Names: dCBT-PF
  Arms: Part 1 - Digital cognitive behavioral therapy; Part 2 - Digital cognitive behavioral therapy

SUMMARY:
The purpose of the study is to assess efficacy and safety of a digital cognitive behavioural therapy for patients with pulmonary fibrosis on anxiety.

DETAILED DESCRIPTION:
Patients will be randomised 1:1 to either receive treatment with the digital therapy, or to act as control group. Patients will be treated for 9 weeks, followed by a 3 week follow-up period. Efficacy will be assessed after 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥22 years at the time of signing the informed consent
2. Self-reported Pulmonary Fibrosis diagnosis
3. A GAD-7 score of ≥5 at pre-screening and baseline
4. If currently on prescribed medication for depression/anxiety, a stable dose for at least 4 weeks prior to baseline
5. CT scan report within 5 years prior to baseline with signs of PF (interstitial changes)
6. Capable of using a mobile device and common applications, and has an appropriate mobile or tablet device

Exclusion Criteria:

1. Self-reported manic disorders, psychotic disorders, schizophrenia, or alcohol/drug abuse during the past 6 months prior to baseline (Visit 1), as judged by the investigator or designee.
2. Self-reported history of hospital admissions due to suicidal behavior or attempts, as judged by the investigator or designee
3. Self-reported previous or current diagnosis of major depressive disorder, as judged by the investigator or designee
4. Verbal and/or written communication problems limiting ability to engage with dCBT-IPF
5. Inability to comply with investigation procedures, due to e.g. cognitive impairment or severe medical conditions as judged by the investigator or designee
6. Currently receiving cognitive behavioral therapy

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2022-04-17 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Horton, MD, Principal Investigator — Curebase study site
Locations (2):
- United States (2):
  - Curebase Study Site, San Francisco, California
  - University of Utah Health, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 subjects were enrolled in the pilot phase (Part 1) to receive 4 weeks of dCBT.
  108 subjects were enrolled in the pivotal phase (Part 2) to recieve either 9 weeks of dCBT or no intervention.
Pre-assignment Details: This investigation consisted of two parts:
  Part 1 - A pilot phase with the key purpose of testing the functionality of dCBT-PF.
  Part 2 - A pivotal phase with the key purpose of evaluating the efficacy of dCBT-PF versus a control on patient-reported psychological symptom burden in patients with PF.
Groups:
- Part 2 - Digital Cognitive Behavioral Therapy: 9 weeks of digital cognitive behavioral therapy.
  Digital cognitive behavioral therapy: Therapy for patients with pulmonary fibrosis
- Part 1 - Digital Cognitive Behavioral Therapy: 4 weeks of digital cognitive behavioral therapy
  Digital cognitive behavioral therapy: Therapy for patients with pulmonary fibrosis
Period: Pilot Investigation - Part 1
Arm/Group | Part 2 - Digital Cognitive Behavioral Therapy | Part 2 - Control Group | Part 1 - Digital Cognitive Behavioral Therapy
Started | 0 (In the pilot phase subjects received 4 weeks digital cognitive behavioral therapy.) | 0 (There was no control group in the Pilot phase) | 11
Completed | 0 | 0 | 10
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Pivotal Investigation - Part 2
Arm/Group | Part 2 - Digital Cognitive Behavioral Therapy | Part 2 - Control Group | Part 1 - Digital Cognitive Behavioral Therapy
Started | 54 | 54 | 0 (Subject from the Part 1 (pilot phase) did not take part in Part 2.)
Completed | 46 | 46 | 0
Not Completed | 8 | 8 | 0
Not completed — Lost to Follow-up | 2 | 2 | 0
Not completed — Withdrawal by Subject | 5 | 2 | 0
Not completed — Death | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Population: One subject randomised to dCBT-PF in Part 2 was not treated, as the subject was unable to download the app.
Groups:
- Part 2 - Digital Cognitive Behavioral Therapy: Part 2: 9 weeks digital cognitive behavioral therapy.
  Digital cognitive behavioral therapy: Therapy for patients with pulmonary fibrosis
- Part 1 - Digital Cognitive Behavioral Therapy: Part 1: 4 weeks digital cognitive behavioral therapy.
  Digital cognitive behavioral therapy: Therapy for patients with pulmonary fibrosis
- Total: Total of all reporting groups
Arm/Group | Part 2 - Digital Cognitive Behavioral Therapy | Part 2 - Control Group | Part 1 - Digital Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 54 | 54 | 11 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (10.21) | 68.9 (8.12) | 71.1 (9.38) | 67.5 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 33 | 5 | 76
  Male | 16 | 21 | 6 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 0 | 5
  Not Hispanic or Latino | 52 | 51 | 11 | 114
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 0 | 6
  White | 49 | 50 | 11 | 110
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1 - Subject Feedback on Functionality and Experience of the dCBT-PF at Week 4
Description: Subject feedback on functionality and experience of the dCBT-PF at Week 4 collected through subject interviews following a separate semi-structured interview guide.
Time Frame: Baseline to Week 4
Population: Qualitative information on functionality and experience was collected from 10 participants.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: 4 Weeks Digital Cognitive Behavioral Therapy.: Digital cognitive behavioral therapy: Therapy for patients with pulmonary fibrosis.
Arm/Group | Part 1: 4 Weeks Digital Cognitive Behavioral Therapy.
Number analyzed (Participants) | 10
Participants
  The device was intuitive and easy to use | 8
  Feature allowing users to review entries in the tool to be added to the device | 2
  Account setting page for users to be added to the device (e.g. for resetting password) | 2
  Difficulties in following the audio tool guidance | 1
  Notifications for daily prompts for device usage to be added | 3

2. Primary Outcome: Part 2 - Change From Baseline in Anxiety Symptom Severity Assessed by Generalized Anxiety Disorder 7-item (GAD-7) at Week 9.
Description: The questionnaire includes 7 questions. Each question will be scored on a 4-point scale from 0 to 3 points. Higher score will mean a worse outcome.
  The GAD-7 represents an anxiety measure based on seven items which are scored from zero to three (0=Not at all,1=Several days, 2=More than half the days and 3=Nearly every day). The composite score can range from 0 to 21 and cut-off scores for mild, moderate and severe anxiety symptoms are 5, 10 and 15 respectively.
Time Frame: Baseline to Week 9
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Digital Cognitive Behavioral Therapy: Part 2: 9 weeks digital cognitive behavioral therapy.
  Digital cognitive behavioral therapy: Therapy for patients with pulmonary fibrosis
- Control Group: No intervention
Arm/Group | Digital Cognitive Behavioral Therapy | Control Group
Number analyzed (Participants) | 54 | 54
score on a scale | -1.8 [-5.9 to 2.4] | 0.9 [-3.3 to 5.1]

3. Secondary Outcome: Part 1 - Safety of dCBT-PF-in Patients With IPF
Description: Information on AEs, ADEs, SAEs, SADE and device deficiencies which could lead to an ADE or SADE was collected at visits at week 2 and week 4.
Time Frame: Baseline to week 4
Population: 1 AE was reported in the pilot phase of the investigation. AE information was not collected for the subject who did not initiate treatment.
Measure: Number; unit: Adverse event
Groups:
- Digital Cognitive Behavioral Therapy: 4 weeks digital cognitive behavioral therapy.
  Digital cognitive behavioral therapy: Therapy for patients with pulmonary fibrosis
Arm/Group | Digital Cognitive Behavioral Therapy
Number analyzed (Participants) | 10
Adverse event | 1

4. Secondary Outcome: Part 2 - Change From Baseline in Anxiety Symptom Severity as Assessed by Hamilton Anxiety Rating Scale (HAM-A) at Week 9
Description: The questionnaire includes 14 questions rating the intensity of psychic and somatic anxiety on a 5-point severity scale. Each item ranging from 0 (not present) to 4 (very severe) will be summed up to give a total possible score of 0 to 56, where lower scores indicate less anxiety.
Time Frame: Baseline to Week 9
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Digital Cognitive Behavioral Therapy | Control Group
Number analyzed (Participants) | 54 | 54
score on a scale | -6.7 [-8.7 to -4.7] | -4.7 [-6.5 to -2.8]

5. Secondary Outcome: Part 2 - Change From Baseline in HRQoL Assessed by King's Brief Interstitial Lung Disease Questionnaire (K-BILD) Psychological Domain Score at Week 9.
Description: The questionnaire includes 3 domains (breathlessness and activities, chest symptoms and psychological). The K-BILD domain and total scores ranges are 0-100; 100 represents the best health status.
Time Frame: Baseline to Week 9
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Digital Cognitive Behavioral Therapy | Control Group
Number analyzed (Participants) | 54 | 54
score on a scale | 8.1 [4.3 to 11.9] | 1.6 [-1.9 to 5.1]

6. Secondary Outcome: Part 2- Change From Baseline in HRQoL Assessed by King's Brief Interstitial Lung Disease Questionnaire (K-BILD) Total Score at Week 9.
Description: as for outcome 5
Time Frame: Baseline to Week 9
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Digital Cognitive Behavioral Therapy | Control Group
Number analyzed (Participants) | 54 | 54
score on a scale | 4.8 [2.3 to 7.3] | 0.4 [-2.0 to 2.9]

ADVERSE EVENTS:
Time Frame: Part 1 - Adverse events/adverse device effects were collected from week 2 until week 4. Subjects were asked at week 2 and 4 if any AE or ADE had been experienced since last visit. AE information was not collected for the subject who did not initiate treatment. Part 2 - Adverse events/adverse device effects were collected from week 3 until week 12. Subjects were asked at week 3, 6, 9 and 12 if any AE or ADE had been experienced since last visit.
Description: In this study, selective AE collection was conducted. All ADE, SAE, or SADE are reported, regardless of treatment-relation. For non-serious, non-treatment-related AEs, only events that were associated with a psychological disorder or with a procedure of the clinical investigation were collected in accordance with the clinical investigation plan and are reported.1 subject in the dCBT-PF arm of Part 2 was randomised but unable to start treatment. AE information was not collected for this subject.
Arm/Group | Part 2 - Digital Cognitive Behavioral Therapy | Part 2 - Control Group | Part 1 - Digital Cognitive Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 1/53 | 4/54 | 0/10
Serious Adverse Events (participants affected / at risk) | 5/53 | 9/54 | 0/10
Other Adverse Events (participants affected / at risk) | 3/53 | 4/54 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 2 - Digital Cognitive Behavioral Therapy (N=53) | Part 2 - Control Group (N=54) | Part 1 - Digital Cognitive Behavioral Therapy (N=10)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 2 - Digital Cognitive Behavioral Therapy (N=53) | Part 2 - Control Group (N=54) | Part 1 - Digital Cognitive Behavioral Therapy (N=10)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 4 (4) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The primary publication should be published by the sponsor prior to any other investigator-initiated publications, manuscripts, abstracts, or presentations.

The results of this clinical investigation may be published or presented at scientific meetings. If this is foreseen, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT05330312/Prot_SAP_000.pdf